CLINICAL TRIAL: NCT01343303
Title: A Double-Blind, Randomized, Placebo-and Active-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-39439335 in Subjects With Osteoarthritis
Brief Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-39439335 in Patients With Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Senior Director, Clinical R&D, Janssen Research & Development, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR018292; 39439335EDI1014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-04-07; First posted 2011-04-28 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, knee; knee pain; pain measurement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Experimental): JNJ-39439335 2 x 5 mg tablets once daily for 21 days
  Interventions: Drug: JNJ-39439335
- 002 (Experimental): JNJ-39439335 2 x 25 mg tablets once daily for 21 days
  Interventions: Drug: JNJ-39439335
- 003 (Other): Naproxen 500 mg capsule every 12 hours for 21 days
  Interventions: Drug: Naproxen
- 004 (Placebo Comparator): Placebo Placebo tablet/capsule every 12 hours for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo tablet/capsule every 12 hours for 21 days
  Arms: 004
Drug: JNJ-39439335 — 2 x 25 mg tablets once daily for 21 days
  Arms: 002
Drug: Naproxen — 500 mg capsule every 12 hours for 21 days
  Arms: 003
Drug: JNJ-39439335 — 2 x 5 mg tablets once daily for 21 days
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the safety of multiple oral doses of JNJ-39439335 and to assess how JNJ-39439335 is absorbed (taken in), distributed, metabolized (broken down), and eliminated from the body (referred to as pharmacokinetics) in osteoarthritis patients. This study will also assess the effectiveness of JNJ-39439335 on pain.

DETAILED DESCRIPTION:
This will be a double-blind (patient and study staff will not know the identity of assigned treatment), randomized (assignment to 1 to 3 treatment groups will be by chance, like "flipping a coin"), placebo-controlled, multiple dose study conducted at up to two clinical sites. Up to 42 patients with osteoarthritis of the knee will be enrolled in 3 cohorts (Cohort 1 to 3). Additional cohorts (up to 14 patients per cohort) may be added after completion of Cohort 3. The study consists of eligibility screening, a treatment phase, and 4 follow-up visits. The study duration for each patient will be approximately 10 weeks. Patients safety will be closely monitored during the study by review of adverse events, electrocardiograms, vital signs (including oral temperature), clinical laboratory tests, and physical examinations. During specified study visits, blood samples will be collected for pharmacokinetics, pharmacodynamics (inpatient patients), and pharmacogenomic (optional) evaluations of JNJ-39439335. The effectiveness of JNJ-39439335 will be evaluated by assessing pain using an 11-point numerical rating scale and by the Western Ontario and McMaster Osteoarthritis Index. In Cohort 1 and 2, all patients will take their study medication orally, twice a day for 21 days. The treatment groups for Cohort 1 are JNJ-39439335 10 mg, naproxen 500 mg every 12 hours, and placebo. The treatment groups for Cohort 2 are JNJ-39439335 25 mg, naproxen 500 mg every 12 hours, and placebo. The treatment groups for Cohort 3 will be determined based on the results of Cohort 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker >= 6 months prior to first dose
* body mass index (BMI) <= 36 kg/m2
* Meet American College of Rheumatology (ACR) clinical classification criteria for osteoarthritis of knee by meeting at least 3 of the following: age > 50, morning stiffness < 30 minutes, crepitus on active motion, bony tenderness, bony enlargement, no palpable warmth of synovium
* Has Functional Class I-III osteoarthritis (OA) of knee with continuing OA-knee joint pain >= 5 days/week x 3 months prior to screening, and has been taking a non-opioid analgesic for OA knee pain daily for >=5 days prior to screening with benefit
* Otherwise healthy based on physical exam, medical history, vital signs, 12-lead electrocardiogram (ECG), can clinical laboratory tests
* Women must be postmenopausal or surgically sterile.

Exclusion Criteria:

* Oral temperature >37.5 deg C at Screening or Day -1
* Failure of burn prevention measures quiz at Screening
* patients with occupations or hobbies in which they are routinely exposed to situations in which they could sustain burns
* orthopedic and/or prosthetic device on target knee joint
* Significant pain outside the target knee, including significant hip or back pain (bilateral knee OA is permitted)
* Unable to discontinue prior analgesic medications/non-steroidal antiinflammatory drugs (NSAIDS) other than paracetamol during the study
* Surgical intervention for any pain within 3 months prior to screening or has plans for surgical intervention while in the study
* History of prior diagnosis of inflammatory arthritis (including rheumatoid arthritis)
* Treatment with local corticosteroid injections or viscosupplementation in target joint, or use of oral or intramuscular corticosteroids, within 3 months prior to Screening
* History of active peptic ulceration, active dyspepsia, gastrointestinal bleeding, Crohn's disease, ulcerative colitis, chronic diarrhea esophageal, and gastric or duodenal ulcer within 3 months prior to screening or any other condition, which in the Investigator's opinion, precludes use of an NSAID.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | From screening up to final follow up visit.
Change from baseline in vital signs, including oral body temperature | From Day -1 up to final follow up visit
Change from baseline in ECG | From Day -1 up to final follow up visit
Change from baseline in clinical laboratory tests | From Day -1 up to final follow up visit
Concentaton of JNJ-39439335 in blood and urine samples | From Day 1 up to final follow up visit
Concentration of JNJ-39439335 in blood and urine samples | From Day 1 up to final follow up visit

SECONDARY OUTCOMES:
Change from baseline in pain numerical rating scale | From Day 2 up to final follow up visit
Change from baseline in Western Ontario and McMaster Osteoarthritis Index (WOMAC) | From Day -1 up to final follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- George, South Africa